CLINICAL TRIAL: NCT06685029
Title: Comparison of Clear Aligner System Produced Directly by the Orthodontist and Indirect Clear Aligner Systems With Fixed Orthodontic Treatment in Terms of Endocrine Disrupting Monomer Release: In-vivo Randomized Controlled Clinical Study
Brief Title: A Comparison of Direct 3D Printed Clear Aligner System and Indirect Clear Aligner Systems With Fixed Orthodontic Treatment in Terms of Endocrine Disrupting Monomer Release, Treatment Effectiveness and Efficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmet Yağcı (Other)
Responsible Party: Sponsor-Investigator, Ahmet Yağcı, PROFESSOR, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDH-2024-13280
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2024-11

CONDITIONS: Endocrine Disruptors
Keywords: Bisphenol A, Clear Aligners, Direct Production.

STUDY DESIGN:
Intervention Model Description: Fifty two patients were divided into 4 groups at study: Group A - Direct In-House Aligner, Group B - Invisalign group, Group C - Clear Correct group, Group D - Fixed Orthodontic Treatment group. Digital models will be obtained from the patients included in study. In addition, saliva samples will be taken at different times of treatment. These saliva samples will be analyzed for Bisphenol A content. The groups will also be compared for the development of white spot lesions. The total treatment time of patients receiving clear aligner treatment and fixed orthodontic treatment will be measured. Treatment effectiveness will be evaluated by scoring digital 3D models taken from patients with the PAR (Peer Assessment Rating) index.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dİrect In-House Aligner Group (Experimental): Patients in this group are treated with clear aligners produced directly by the clinician. The physical model production step is eliminated with direct production technique.Intraoral scan images were obtained from these patients with the 3Shape TRIOS (3Shape, Copenhagen, Denmark) scanning device. Then, the 3D scan images were transferred to the Maestro 3D Dental Studio (New Age, Pisa, Italy) computer software. Using these scan images, the teeth were gradually moved according to the planned final treatment result. The number of clear paligners required is calculated by the program according to the total amount of planned tooth movement. Then, Tera Harz TC-85DAC (Graphy, Seoul, Korea) resin and Asiga MAX UV (Asiga, Sydney, Australia) 3D printer were used for the direct production of the plates designed in the program. The aligners produced were then delivered to the patients.
  Interventions: Device: Clear aligner treatment
- Invisalign Group (Experimental): Intraoral scan images were obtained with the 3Shape TRIOS (3Shape, Copenhagen, Denmark) scanning device from patients who would receive Invisalign (Align Technology, Santa Clara, CA) clear aligners. These 3D intraoral scan images, together with the intraoral and extraoral photographs, radiographic records, and clinical examination findings obtained from the patients, were uploaded to the cloud software 'ClinCheck' for Invisalign . Necessary instructions were written regarding the patients' treatment plans. Afterwards, patient specific 3D treatment simulations sent to the clinician by the companies were reviewed and the necessary revisions were made. The final accepted treatment plan was approved and the aligners were produced by the relevant companies and sent to the clinic.The clear aligners produced are delivered to the patients and treatment started.
  Interventions: Device: Clear aligner treatment
- ClearCorrect Group (Experimental): Intraoral scan images were obtained with the 3Shape TRIOS (3Shape, Copenhagen, Denmark) scanning device from patients who would receive Invisalign (Align Technology, Santa Clara, CA) and ClearCorrect (ClearCorrect®, Round Rock, TX, USA) clear aligners. These 3D intraoral scan images, together with the intraoral and extraoral photographs, radiographic records, and clinical examination findings obtained from the patients, were uploaded to the cloud software 'ClinCheck' for Invisalign . Necessary instructions were written regarding the patients' treatment plans. Afterwards, patient specific 3D treatment simulations sent to the clinician by the companies were reviewed and the necessary revisions were made. The final accepted treatment plan was approved and the aligners were produced by the relevant companies and sent to the clinic.The clear aligners produced are delivered to the patients and treatment started.
  Interventions: Device: Clear aligner treatment
- Fixed Orthodontic Treatment Group (Experimental): In the fixed orthodontic treatment group, all tooth surfaces to which brackets would be bonded were etched with 37% phosphoric acid (dline Phosphoric Acid Etching Gel UAB, Medicinos linij Karaliauciaus str. 29 LT-78348 Siauliai Lithuania) for 30 seconds, then bond (3M Unitek Transbond XT, Minnesota, U.S.A.) was applied and light was applied to all teeth separately for 5 seconds with a light device (Valo Cordless curing light Ultradent Products, Inc. 505 W. Ultradent Drive (10200 South) South Jordan, UT 84095) [165, 166]. Afterwards, composite (3M Unitek Transbond XT, Minnesota, U.S.A.) was applied to the base of the metal brackets (AO Mini Master Roth 018, Altenhofstrasse 80, 66386 St. Ingbert, Germany) and after it was placed on the tooth surface and the composite residues around the bracket were cleaned, light was applied for 5 seconds for each bracket. Then, arch wires were applied and the fixed orthodontic treatment of the patients was started.
  Interventions: Device: Fixed Orthodontic Appliance Treatment

INTERVENTIONS:
Device: Clear aligner treatment — Clear aligners are appliances that allow the teeth to be gradually moved to the desired final position, as planned in the computer program, in a way that each aligner will perform a part of the total movement with its use.
  Arms: ClearCorrect Group; Dİrect In-House Aligner Group; Invisalign Group
Device: Fixed Orthodontic Appliance Treatment — Fixed orthodontic treatment is a type of orthodontic treatment performed by applying brackets and wires to the teeth and is considered the gold standard for orthodontic treatments.
  Arms: Fixed Orthodontic Treatment Group

SUMMARY:
The aim of this study is to evaluate the release of endocrine disrupting monomers from clear aligners as a result of exposure to intraoral factors by measuring their concentration in saliva and to evaluate their reliability of use in terms of general health by comparing them with the fixed orthodontic treatment group. It is also aimed to compare the groups in terms of treatment effectiveness and efficiency.

DETAILED DESCRIPTION:
The aim of our study is to evaluate the saliva concentration of endocrine-disrupting monomers released from attachments used and clear aligners produced directly by the orthodontist in the clinic and indirectly produced by companies. Accordingly comparing them with the fixed orthodontic treatment group and assessing clear aligner's safety for general health. It is also aimed to compare the groups in terms of treatment effectivenes and total time spent . Endocrine-disrupting chemicals are substances that interfere with the synthesis, metabolism, or effects of hormones, causing deviation from normal reproduction and homeostatic control in organisms. Bisphenol A (BPA), a monomer, is also included in the chemicals listed as endocrine disruptors by the World Health Organization. Different studies have suggested that Bisphenol A may cause adverse health effects by acting as an endocrine disruptor. While previous research has been conducted on BPA release or monomer leakage related to orthodontic materials, there is limited evidence regarding the safety aspects of thermoplastic aligners or retainers. The concentrations of endocrine-disrupting monomers in the saliva of patients undergoing treatment with directly produced aligners by orthodontists and indirectly produced aligners by companies will be examined in comparison to patients undergoing fixed orthodontic treatment. Patients will not receive any treatment other than routine orthodontic care.

ELIGIBILITY:
Inclusion Criteria:

* Absence of primary teeth in the oral cavity, with permanent teeth fully erupted,
* Presence of a non-extraction orthodontic treatment plan,
* Age range of 15 to 24 years,
* Presence of mild to moderate dental crowding (0-6 mm of crowding),
* Classification as skeletal Class I (ANB: 2±2°),
* Absence of any craniofacial anomalies,
* Normal vertical growth pattern (Sn-GoGn: 32±6°),
* No congenital tooth agenesis (excluding third molars),
* Absence of atypical tooth morphology,
* No extracted permanent teeth,
* Absence of dental caries,
* Good level of oral hygiene,
* Healthy periodontal tissues.

Exclusion Criteria:

* Presence of any systemic disease,
* History of previous fixed orthodontic treatment,
* History of allergy to any dental material,
* Use of medications containing estrogen analogs,
* Patients with a history of xerostomia and a salivary flow rate of less than 0.1 ml per minute,
* Patients with more than five composite restorations.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Bisphenol A Concentration | up to 1 year
  Bisphenol A concentration in patients' saliva is measured as ng/ml.

SECONDARY OUTCOMES:
Treatment efficiency | up to 1 year
  The total time required to complete the treatment is calculated.
Treatment Effectiveness (via PAR İndex) | up to 1 year
  The percentage decrease in the PAR score is calculated for each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University,Faculty of Dentistry,Department of Orthodontics, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kassam SK, Stoops FR. Are clear aligners as effective as conventional fixed appliances? Evid Based Dent. 2020 Mar;21(1):30-31. doi: 10.1038/s41432-020-0079-5. PMID 32221494
- [Background] Iliadi A, Koletsi D, Papageorgiou SN, Eliades T. Safety Considerations for Thermoplastic-Type Appliances Used as Orthodontic Aligners or Retainers. A Systematic Review and Meta-Analysis of Clinical and In-Vitro Research. Materials (Basel). 2020 Apr 14;13(8):1843. doi: 10.3390/ma13081843. PMID 32295303
- [Background] Raghavan AS, Pottipalli Sathyanarayana H, Kailasam V, Padmanabhan S. Comparative evaluation of salivary bisphenol A levels in patients wearing vacuum-formed and Hawley retainers: An in-vivo study. Am J Orthod Dentofacial Orthop. 2017 Mar;151(3):471-476. doi: 10.1016/j.ajodo.2016.07.022. PMID 28257731
- [Background] Yazdi M, Daryanavard H, Ashtiani AH, Moradinejad M, Rakhshan V. A systematic review of biocompatibility and safety of orthodontic clear aligners and transparent vacuum-formed thermoplastic retainers: Bisphenol-A release, adverse effects, cytotoxicity, and estrogenic effects. Dent Res J (Isfahan). 2023 Mar 28;20:41. eCollection 2023. PMID 37180685